CLINICAL TRIAL: NCT06922409
Title: The Effects of Naturalistic Light on Post Stroke Complications Related Brain Areas in Stroke Patients During Admission for Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Chromaviso A/S (Other)
Responsible Party: Principal Investigator, Anders Sode West, MD, Ph.D. Principal Investigator, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-22014644
Record Dates: First submitted 2025-03-27; First posted 2025-04-10 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Post Stroke Depression; Post Stroke Fatigue; Circadian Dysregulation; Stroke
Keywords: circadian rhythm disruption; Stroke; Post Stroke Depression; Post Stroke Fatigue; Light therapy; Circadian Light
MeSH Terms: conditions — Chronobiology Disorders; Stroke

STUDY DESIGN:
Intervention Model Description: Study Design:
  Case-control study
  Study description:
  Patients admitted at the acute stroke unit will be screened for fatigue and depression. The patients will be selected for the study by the present and absent of moderate-severe depression and fatigue (50%+50%). The control group will be patients without any symptoms of depression and fatigue. The intervention group will be patients scored to have moderate-severe depression and fatigue. All patients must be selected to neurorehabilitation for a minimum of 10 days where the intervention (naturalistic light) is installed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate-severe depression or/and fatigue (Active Comparator): Naturalistic Light Intervention
  Interventions: Device: Naturalistic Light Intervention
- No measured depression or/and fatigue (Active Comparator): Naturalistic Light Intervention
  Interventions: Device: Naturalistic Light Intervention

INTERVENTIONS:
Device: Naturalistic Light Intervention — Naturalistic light as an Intervention A 24-hour naturalistic lighting scheme is implemented in all areas and rooms in the unit at Rigshospitalet Glostrup with a computer-controlled lighting scheme (ChromaViso, Denmark). The naturalistic lighting scheme is constantly running. The lighting imitate the sunlight rhythm following the principles of Lucas et al.
  Other Names: Circadiain Light Intervention; Dynamic Light Intervention

SUMMARY:
Background:

Light is the most important regulator of circadian rhythm. Naturalistic light, which contains the spectrum of sunlight throughout the day, has been shown to have a positive impact on mental states such as depression and fatigue in stroke and other diseases requiring long-term hospitalization.

Depression and fatigue are very common complications after stroke, with a frequency of 30% and 85%, respectively. Both are significantly related to reduced quality of life and early death. Both the causes and pathophysiology behind these complications are unknown, but it is assumed that disturbances (inflammation and cell death) in brain areas and brain networks related to arousal, sleep, circadian rhythm, and the frontal lobe play a role.

The hypothesis is that it is possible to detect changes in brain networks related to depression and fatigue by MRI, and that naturalistic light will affect these changes.

Method:

Stroke patients requiring a minimum of 10 days of rehabilitation are transferred to a neurorehabilitation unit with naturalistic lighting.

Examination:

Validated tests for fatigue, depression, sleep and cognitive functions.

Pathophysiological studies:

* MRI focusing on cerebral blood flow, metabolism, and cerebral networks.
* Spinal fluid analyses for hormones and markers involved in immunological response as well as wakefulness/arousal and depression.
* Sleep assessments.

DETAILED DESCRIPTION:
OBJECTIVE AND PURPOSE

To investigate the effect of naturalistic lighting (i.e., artificial light imitating the sunlight rhythm and spectrum) on depression, sleep, executive cognition, and fatigue in a hospital setting among patients admitted for post-stroke rehabilitation. The effect is planned to be measured by questionnaires, MRI modalities, and CSV markers for localizing inflammation, levels of hypocretin and sleep. The hypothesis is based on the findings from the previously light trial.

BACKGROUND INFORMATION

Stroke annually affects approximately 12,000 Danes and there are approximately 75,000 stroke survivors with sequelae after stroke. Stroke is the major cause of acquired cerebral disability among adults, the second most common cause of dementia and the fourth leading cause of death. An effective rehabilitation program is mandatory for optimal recovery; however, post stroke complications in relation to circadian rhythm disruptions counteracts this.

The circadian rhythm association The circadian response is especially sensitive of short-wavelength blue light because of the blue light-sensitive photopigment Melanopsin in the retina, which communicates with the suprachiasmatic nucleus (SCN) through the retinohypothalamic tract (RHT). As sunlight contains blue light, it is essential to imitate the stimulation during the day to entrain the circadian rhythm. Active, working people are exposed to bright sunlight during the day to regulate their circadian rhythm but in hospitals, rehabilitation patients are often indoors and receive only bright light through the hospital window and disturbing light in night time by normal light bulbs.

The previously light trial A light trial was conducted in 2014-2015 with the title "The effect of naturalistic light in stroke patients" (Danish scientific ethics committee (H-4-2013-114) and the Danish Data Protection Agency (2007-58-0015). ClinicalTrials.gov Identifier: NCT02186392.). The study was a large project investigating the effect of naturalistic light on human health measured by psychological parameters, biochemical parameters, fatigue and sleep.

The trial was carried out in the Stroke Rehabilitation unit, Department of Neurology, Rigshospitalet, Copenhagen. The study was a randomized controlled study with two arms. Stroke patients at the acute stroke unit were randomized to either an intervention rehabilitation unit (IU) equipped with naturalistic lighting or a control rehabilitation unit (CU) with standard lighting.

One of the main findings was a significant decrease depressive mood by 51.9%, decreased fatigue by 20.6%, decreased anxiety by 28,6%, increased rested feeling by 41,6% and increased well-being by 46,5%. Furthermore, the study found increased serum cortisol morning levels and increased levels of melatonin and rhythmicity in patients exposed to naturalistic light during admission. No difference in cognition, sleepiness and sleep quality were detected. In papers that are currently undergoing peer-review have showed disturbed endocrinological parameters after stroke, but no effect of the naturalistic light indicating that light may be a central circadian regulator.

Light and depression A proximately one third of stroke patients (30-50%) suffer of Post Stroke Depression (PSD). PSD has been significantly associated with increased mortality approx. 50%, taking risk factors into account. The mortality is reduced to 20% by treatment vs 65% without treatment. PSD is also associated to new stroke incidence, reduced participation in rehabilitation (54%), reduced cognitive function, double the number of suicides, increased use of health services and decreased activity of daily living.

The circadian rhythm is responsible for the circadian expression and activity of several neurotransmitters and circadian-controlled genes known as clock genes.

Based on our previous results and the literature, naturalistic light appears to reduce the depressive mood in the post stroke brain. However, the pathophysiology of PSD is still unclear and there is still no clear evidence linking brain lesions to PSD. Therefore, investigating cerebral serotonin transporter binding, the brains activity and functional network connectivity, especially output from SCN, measured by brain scans may obtain knowledge about the source of the PSD.

Post Stroke Fatigue Post stroke fatigue (PSF) is defined by extreme tiredness resulting from mental or physical exertion or illness and affect 25% to 85% of stroke patients (75% in the previously described light study). PSF reported by forty percent of stroke patients to be the worst or one of the worst sequelae after stroke.

Complications after PSF, has been correlated with the following: reduced functional outcome, decrease in activities of daily living (ADL) and mortality.

The pathophysiological and anatomical explanation behind PSF is like PSD not fully understood. However, brain structures that have been found to be significantly associated to PSF are the thalamus, brainstem, subcortical region and basal ganglia which are known to have connections to the SCN, why SCN may be an important stimulator.

Cognitive executive functions The prevalence of post stroke cognitive impairment varies between studies but range from 7.5% to 72%. It has been proven that the cognitive function in humans becomes impaired with disturbance of the circadian rhythm. The physiology behind circadian disturbance and cognitive dysfunction is not completely known, but brain regions outside of the SCN may be part of the mechanism where Diffusion tensor tractography (DTT) appear to visualize the structures.

In relation to the above, cerebral hypoperfusion may also be relevant to examine as reduced cognition, like depression, has been correlated to regional cerebral hypoperfusion.

Naturalistic light as an Intervention A 24-hour naturalistic lighting scheme is already implemented in all areas and rooms in unit N35 at Rigshospitalet Glostrup with a computer-controlled lighting scheme (ChromaViso, Denmark). The naturalistic lighting scheme is constantly running.

METHOD

Experimental participants and the Intervention during hospitalization The intervention group and the control group are stroke patients admitted to the acute stroke unit and considered suitable for admission in the rehabilitation's unit, Department of Neurology, Rigshospitalet Glostrup during the period February 1th 2025 to February 1th 2027.

Patients admitted at the acute stroke unit will be screened for fatigue and depression. The patients will be selected for the study by the present and absent of moderate-severe depression and fatigue (50%+50%). The control group will be patients without any symptoms of depression and fatigue. The intervention group will be patients scored to have moderate-severe depression and fatigue. All patients must be selected to neurorehabilitation in our rehabilitation unit for a minimum of 10 days which include rehabilitation through physiotherapy, occupational therapist, speech therapist or a neuropsychologist. The rehabilitation unit is the intervention unit where the Naturalistic light is installed. In the acute stroke unit, the patient receives the normal initial assessment, blood samples, physical neurological somatic examination, and the paraclinical examination program after stroke.

At the inclusion, patients will be assessed by the following assessments mentioned below, which again will be evaluated at discharge.

The numbers of patients who are expected to be included in total are 45 patients, which is estimated to be 42 enrolled and completed patients after dropout (i.e. 21 patients in each group). In addition, same makers from blood and CSF will be collected from 10 healthy subjects.

Trial Design Case-control study with two arms. The number of patients who are expected to be included are 45.

Assessments

1. Stroke classification scales
2. Questionnaires and physiological tests of sleep quality
3. Questionnaires for depression
4. Test for executive cognitive function performed by neuropsychologist
5. Test for fatigue
6. Testing for mobilization level and status of physical rehabilitation
7. Cerebrospinal fluid (CSF): Special inflammation makers, Neuronal injury and neurotransmitters in relation to sleep and depression.
8. MRI perfusion and network sequences

STATISTICS

Power and sample size analysis 5% cut-off point.

Depression and Fatigue:

Experience from our previous trials, we estimate that at least 40 patients must be included regarding the Multidimensional Fatigue Inventory (MFI-20) and Major depression inventory test (MDI).

MRI:

The power calculation is based on literature using different toolboxes for MRI power calculations e.g www.neuropowertools.org. With a 5% cut-off point and power on 80% up against various test for multiple testing, must the included number of subjects be above 40.

Sleepiness and sleep quality:

It was not possible to detect any significance in our previously trial. However, the lack of significance may also be related to the patent cohort due to impaired sleep network as a result of the stroke, why a significant outcome may be found in subgroups and therefore not a power problem in this trail.

ELIGIBILITY:
Inclusion Criteria:

* Patients scoring moderate-severe fatigue and/or depression OR NO fatigue and/or depressione which are evaluated as candidates for the rehabilitation unit.

Exclusion Criteria:

* GCS < 15
* No functioning nervus opticus or retina in both eyes
* Unable to open both eyes
* Non communicating patients e.g. severe aphasia (incompetent patients)
* Unable to cooperate to the physical examinations
* Less than 10 days of hospitalization in the rehabilitation department
* Claustrophobia
* If the sub investigator finds the study participant unfit to conduct the investigations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue and depression | From admission at the rehabilitation unit to the time of discharge aprox. 10 days.
  Primary hypothesis: Naturalistic light reduce the major depression inventory questionnaire score and multidimensional fatigue inventory questionnaire score from baseline til discharge. Mood-related network will too show positive changes measured by whole brain resting-state connectivity in post-stroke patients compared with a control group without fatigue and depression.

SECONDARY OUTCOMES:
Cognitive function | From admission to the neurorehabilitation unit to the time of discharge aprox 10 days..
  Secondary hypothesis: Naturalistic light improves executive cognitive function and processing speed in test included in the Neuropsychology assessments (Verbal fluency, 1 minute each per test: Category fluency (animals) and lexical fluency (s words and a words), System Digit Modalities Test (SDMT), and Stroop test) and furthermore modifies cognitive related network activation measured by fMRI in post-stroke patients compared with a control group without cognitive impairment.
Sleep quality | From admission to the neurorehabilitation unit to the time of discharge aprox. 10 days..
  Secondary hypothesis: Naturalistic light improves sleep quality from baseline to discharge measured by polysomnography and Pittsburgh Sleep Quality Index questionnaire in post-stroke patients compared with a control group without poor sleep quality.
Hypocretin | From admission to the neurorehabilitation unit to the time of discharge aprox. 10 days..
  Secondary hypothesis: Naturalistic light increase hypocretin levels from baseline to discharge in post stroke patients with measured fatigue and sleepiness compared to a control group without fatigue and sleepiness.
CFS inflammation | From admission to the neurorehabilitation unit to the time of discharge aprox. 10 days.
  Secondary hypothesis: The severity of post stroke fatigue and post stroke depression is associated to the level of markers related to cerebral inflammation based on measured CFS inflammation and naturalistic light will decrease this inflammation compared to a control group without fatigue and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Sode West, MD, PhD, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Faculty of Health and Medical Sciences - University of Copenhagen, Glostrup Municipality, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
The confidentiality of this data is not yet known.

REFERENCES:
- [Background] West A, Jennum P, Simonsen SA, Sander B, Pavlova M, Iversen HK. Impact of naturalistic lighting on hospitalized stroke patients in a rehabilitation unit: Design and measurement. Chronobiol Int. 2017;34(6):687-697. doi: 10.1080/07420528.2017.1314300. Epub 2017 Apr 21. PMID 28430522